CLINICAL TRIAL: NCT01752205
Title: A Randomized Phase III Study: Paclitaxel Plus Radiation Therapy With or Without Erlotinib in Treating Patients With Esophageal Squamous Carcinoma
Brief Title: Paclitaxel Plus Radiation With Erlotinib to Treat Esophageal Squamous Carcinoma
Acronym: ESCC-307PLAH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Responsible Party: Principal Investigator, Xu jianming, The Affiliated Hospital of the Chinese Academy of Military Medical Sciences, The Affiliated Hospital of the Chinese Academy of Military Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESCC-307PLAH-XJM
Record Dates: First submitted 2012-12-16; First posted 2012-12-19 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Esophageal Squamous Carcinoma
Keywords: Esophageal Squamous Carcinoma; Erlotinib; Chemoradiotherapy
MeSH Terms: interventions — Paclitaxel; Erlotinib Hydrochloride; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemoradiotherapy (Active Comparator): The patients will receive radiation therapy QD, 5 days a week and receive paclitaxel IV ，dosing schedule: 45mg/m2/w.
  Interventions: Drug: Paclitaxel; Radiation: Radiation therapy
- Erlotinib and chemoradiotherapy (Experimental): The patients will receive radiation therapy QD, 5 days a week and receive paclitaxel IV (45mg/m2/w) and erlotinib PO QD.
  Interventions: Drug: Paclitaxel; Drug: Erlotinib; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Paclitaxel — 45mg/m2/w,total 6 weeks
Drug: Erlotinib — 150mg/d,days 1-42,total 6 weeks
  Arms: Erlotinib and chemoradiotherapy
Radiation: Radiation therapy
  Other Names: radiation therapy QD, 5 days a week,95%PTV 60Gy/2Gy/30f,total 6 weeks

SUMMARY:
The purpose of this study is to test the safety and effectiveness of erlotinib and chemoradiotherapy in patients with unresectable esophageal or gastro-esophageal squamous cancer .

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed squamous cell carcinoma of esophagus or Esophagogastric Junction
2. Age >= 18
3. ECOG PS 0-2
4. Ineligibility for surgery
5. No prior palliative therapy
6. At least one bidimensionally measurable disease as defined by RECIST ver 1.1
7. Adequate organ function for treatment

   * Absolute neutrophil count (ANC)>=1000cells/mm3
   * Platelets >=100000 cells/mm3
   * Estimated creatinine clearance>=50mL/min, or serum creatinine<1.5 x institution upper limit of normal
   * Bilirubin=<1.5 x upper limit of normal(ULN)
   * AST(SGOT)=<2.5 x ULN (5.0xULN if hepatic metastases)
   * ALT(SGPT)=<2.5 x ULN (5.0xULN if hepatic metastases)
   * 12-Lead electrocardiogram(ECG) with normal tracing or non-clinically significant changes that do not require medical intervention
   * QTc interval =<470 msec and without history of Torsades de Points or other symptomatic QTc abnormality
   * LVEF (by MUGA or echocardiogram) of >=50%.
8. The patient has provided signed informed consent and is amenable to compliance with protocol schedules and testing.

Exclusion Criteria:

1. Previous treatment with small molecule EGFR tyrosine kinase inhibitors
2. Any major operation within 4 weeks of baseline disease assessment
3. Any clinically significant gastrointestinal abnormalities which may impair intake or absorption of the study drug
4. CNS metastasis with continuous corticosteroid use within 4 weeks of baseline disease assessment
5. Patients with known interstitial lung disease
6. Patients with uncontrolled or significant cardiovascular disease (AMI within 12 months,Unstable angina within 6 months, NYHA Class III, IV Congestive heart failure or left ventricular ejection fraction below local institutional lower limit of normal or below 45%, Congenital long QT syndrome, Any significant ventricular arrhythmia, Any uncontrolled second or third degree heart block, Uncontrolled hypertension)
7. Previous or concurrent malignancy except for basal or squamous cell skin cancer and/or in situ carcinoma of the cervix, or other solid tumors treated curatively and without evidence of recurrence for at least 5 years prior to study entry.
8. Pregnant or breast-feeding women
9. Other severe acute or chronic medical condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the patient inappropriate for entry into this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-05 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 2 year

SECONDARY OUTCOMES:
Tumor response rate | 1 year
disease control rate | 1 year
overall survival | 5 year
adverse events | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Xu jianming, M.D., Principal Investigator — The Affiliated Hospital of the Chinese Academy of Military Medical Science
Locations (1):
- 307 Hospital of PLA, Beijing, Beijing Municipality, China